CLINICAL TRIAL: NCT05266859
Title: Comparison of Efficacy of Platelet-rich Fibrin, Mineral Trioxide Aggregate and Calcium Hydroxide as Pulpotomy Medicaments in Permanent Teeth With Irreversible Pulpitis
Brief Title: Efficacy of PRF and MTA as Compared to Calcium Hydroxide for Pulpotomy in Human Irreversibly Inflamed Permanent Teeth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Liaquat College of Medicine and Dentistry (Other)
Collaborators: Ziauddin University (Other)
Responsible Party: Principal Investigator, Naheed Najmi, Vice Principal and Registrar, Liaquat College of Medicine and Dentistry
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC/13/17
Record Dates: First submitted 2022-02-18; First posted 2022-03-04 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Pulpitis - Irreversible; Tooth Decay
Keywords: MTA; Calcium Hydroxide; PRF; Pulpotomy; Irreversible pulpitis; Permanent teeth; Medicament
MeSH Terms: conditions — Dental Caries | interventions — Calcium Hydroxide; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I- Calcium hydroxide (Control) (Active Comparator): Group I will receive Calcium hydroxide . Calcium hydroxide is a gold standard medicament for the pulpotomy in deciduous teeth. It has antibacterial effects and widely used to disinfect the root canals.
  This group will act as a control
  Interventions: Other: Calcium hydroxide
- Group II- MTA (Experimental) (Experimental): Group II will receive MTA (Mineral Trioxide Aggregate). MTA is a calcium silicate based highly biocompatible material that is commonly used for pulpotomies in deciduous teeth along with the regenerative procedures in permanent and deciduous teeth
  Interventions: Other: MTA
- Group III- PRF (Experimental) (Experimental): Group III will receive PRF. PRF is platelet-rich fibrin that is a biocompatible product derived from patient's own blood. It is formed by centrifugation of the blood of the patient. It provides the growth factors and promotes regeneration of the pulp
  Interventions: Other: PRF

INTERVENTIONS:
Other: Calcium hydroxide — Calcium hydroxide in the power/liquid form will be used and placed on the exposed pulp
  Arms: Group I- Calcium hydroxide (Control)
Other: MTA — Mineral trioxide aggregate will be used as a powder / liquid form and placed over the exposed pulp
  Arms: Group II- MTA (Experimental)
Other: PRF — PRF will be placed directly over the exposed pulp
  Arms: Group III- PRF (Experimental)

SUMMARY:
Of all the various pulpotomy medicaments that have been studied till to date, three agents have been selected for this study to compare their efficacy. CH being the control, MTA being one of the most recommended biomaterial and PRF that in addition to being a biomaterial is an autologous agent. Uptil now there have been no prospective trials using these three pulpotomy agents in mature permanent teeth with irreversible pulpitis in our part of the world and even the international studies that have been done utilized different methodologies with no unanimous conclusion. This is the reason that at present this treatment regime (pulpotomy) showing better perspectives cannot be presented with confidence as a predictable treatment option to the patients with irreversible pulpitis. By virtue of this study this challenge is being undertaken.

Hypothesis:

ALTERNATE HYPOTHESIS There is a difference between the efficacy of the PRF, MTA and CH when used as pulpotomy medicaments in mature permanent teeth with irreversible pulpitis NULL HPOTHESIS There is no difference in efficacy of the PRF, MTA and CH when used as pulpotomy medicaments in mature permanent teeth with irreversible pulpitis

ELIGIBILITY:
Inclusion Criteria:

* Patients with permanent teeth with completely formed roots diagnosed with irreversible pulpitis i.e. showing signs and symptoms as spontaneous, lingering pain initiated by hot and cold stimulus and /or radiating. Pulp being exposed or near to exposure by caries or alternatively by trauma.

Exclusion Criteria:

* CLINICALLY Teeth with

  * Necrotic pulp
  * History of swelling, abscess , fistula and/ or sinus tract
  * Doubtful restorability as indicated by over all Dental Practicality Index- (DPI) > 2 (Dawood and Patel 2017) will be excluded
  * Periodontal disease
  * Uncontrolled bleeding (more that 10 mins.) of pulp after removal of inflamed part.
  * No bleeding of pulp at all after access into pulp RADIOGRAPHICALLY (with the use of periapical radiographs) Teeth with
  * Internal/ external pathologic root resorption
  * Pulp canal obliteration
  * Periapical / furcal radiolucency
  * Resorbed roots.
  * Crestal bone loss Generally patients
  * With systemic diseases, bleeding disorders, physical or mental disability, pregnant or nursing.
  * On opioid or steroid therapy or anticoagulants and/or on any kind of antibiotics.
  * Who have gone through some previous treatment for the same tooth other than filling.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Clinical Success or Failure | 12 months
  Incidence of pain, swelling, sinus tract formation, tenderness to percussion after specified time period after intervention
Radiographic Success or Failure | 12 months
  Incidence of Periapical radiolucency or widening and Resorption

CONTACTS AND LOCATIONS:
Locations (1):
- Liaquat College of Medicine and Dentistry, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No